CLINICAL TRIAL: NCT00145496
Title: A Multicenter, Double-Blind, Flexible -Dose, 6-Month Trial Comparing the Efficacy and Safety of Asenapine With Olanzapine in Stable Subjects With Predominant, Persistent Negative Symptoms of Schizophrenia.
Brief Title: Efficacy and Safety of Asenapine Compared With Olanzapine in Patients With Persistent Negative Symptoms of Schizophrenia (A7501013)(COMPLETED)(P05771)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05771; Aphrodite; A7501013
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Results first posted 2010-03-25 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — asenapine; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- asenapine (Experimental)
  Interventions: Drug: Asenapine
- olanzapine (Active Comparator)
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Asenapine — 5-10 mg sublingually twice daily for up to 26 weeks
  Arms: asenapine
Drug: Olanzapine — 5-20 mg by mouth once daily for up to 26 weeks
  Arms: olanzapine

SUMMARY:
Treatment with conventional antipsychotics such as haloperidol has little effect or may sometimes even worsen negative symptoms (such as blunted affect, emotional withdrawal, and poor rapport) of schizophrenia. The newer "atypical" antipsychotics agents, such as olanzapine, has shown improvement in the treatment of negative symptoms in acute trials. The purpose of this study is to compare an investigational compound (asenapine) with a marketed agent (olanzapine) in the treatment of stable subjects with persistent negative symptoms of schizophrenia for 6 months. Patients completing this study may be eligible to participate in an extension 6 months of treatment. Patients are required to have stable symptoms prior to entry into study.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented current diagnosis of schizophrenia of paranoid, disorganized, catatonic, residual, or undifferentiated subtype with persistent negative symptoms.
* No increase in level of psychiatric care during the past few months due to worsening of symptoms of schizophrenia.
* Caregiver required.

Exclusion Criteria:

* Have an uncontrolled, unstable clinically significant medical condition.
* Have any other psychiatric disorder other than schizophrenia as a primary diagnosis including depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2004-12; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

REFERENCES:
- [Result] Buchanan RW, Panagides J, Zhao J, Phiri P, den Hollander W, Ha X, Kouassi A, Alphs L, Schooler N, Szegedi A, Cazorla P. Asenapine versus olanzapine in people with persistent negative symptoms of schizophrenia. J Clin Psychopharmacol. 2012 Feb;32(1):36-45. doi: 10.1097/JCP.0b013e31823f880a. PMID 22198451

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Asenapine | Olanzapine
Started | 244 (Subjects who received randomized treatment assignment and at least one dose of study medication.) | 224 (Subjects who received randomized treatment assignment and at least one dose of study medication.)
Completed | 121 | 143
Not Completed | 123 | 81
Not completed — Adverse Event | 42 | 30
Not completed — Lack of Efficacy | 12 | 7
Not completed — Withdrawal by Subject | 32 | 26
Not completed — Lost to Follow-up | 12 | 5
Not completed — Other | 25 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asenapine | Olanzapine | Total
Number analyzed (Participants) | 244 | 224 | 468
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (11.43) | 42.8 (11.27) | 42.9 (11.34)
Age, Customized [Number; unit: participants]
  <18 years | 0 | 0 | 0
  18 to 64 years | 239 | 217 | 456
  >=65 years | 5 | 7 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 54 | 122
  Male | 176 | 170 | 346
Body Weight [Mean (Standard Deviation); unit: kg] | 84.0 (19.01) | 85.7 (18.71) | 84.8 (18.86)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Negative Symptoms of Schizophrenia Measured by the Negative Symptom Assessment (NSA) Scale Total Score
Description: The NSA Scale is a 16-item clinician-rated instrument for rating the negative symptomatology of schizophrenia. Total score ranges from 16 to 96, with greater scores indicating greater severity of symptoms.
Time Frame: Day 182
Population: Analysis was intent to treat - subjects who received at least 1 dose of double-blind trial medication and had at least 1 post-baseline value.
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Asenapine | Olanzapine
Number analyzed (Participants) | 234 | 218
Units on a Scale
  Baseline | 60.4 (0.80) | 61.3 (0.80)
  Change From Baseline at Day 182 | -9.7 (0.95) | -9.2 (0.89)
Statistical Analysis 1: Comparison: Asenapine vs Olanzapine; The null hypothesis was that there was no difference in change from baseline in NSA Scale total score between asenapine and olanzapine at Day 182; Test type: Superiority or Other; p = 0.7177, Mixed Model for Repeated Measurements — The test of hypothesis was a 2-tailed test with alpha=0.05 (0.049 to adjust for one interim analysis)

2. Secondary Outcome: Change From Baseline in Quality of Life Measured by the Quality of Life Scale (QLS) Total Score
Description: The Quality of Life Scale is a 21-item clinician-rated scale for rating psychosocial functioning (Interpersonal Relations, Instrumental Role, Intrapsychic Foundations, and Common Objects and Activities). The score ranges from 0 to 126, with greater values indicating better quality of life.
Time Frame: Day 182
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Asenapine | Olanzapine
Number analyzed (Participants) | 234 | 218
Units on a Scale
  Baseline | 46.3 (1.20) | 44.2 (1.20)
  Change From Baseline at Day 182 | 11.1 (1.54) | 7.1 (1.41)
Statistical Analysis 1: Comparison: Asenapine vs Olanzapine; The null hypothesis was that there was no difference in change from baseline in QLS total score between asenapine and olanzapine at Day 182; Test type: Superiority or Other; p = 0.0565, Mixed Model for Repeated Measurements — The test of hypothesis was a 2-tailed test with alpha=0.025 nominal significance using the Bonferroni adjustment to account for multiplicity of the key secondary comparisons

3. Secondary Outcome: Change From Baseline in Body Weight
Time Frame: Day 182
Population: as for outcome 1
Measure: Mean (Standard Error); unit: kg
Arm/Group | Asenapine | Olanzapine
Number analyzed (Participants) | 234 | 218
kg
  Baseline | 84.2 (1.40) | 84.7 (1.40)
  Change From Baseline at Day 182 | 0.0 (0.43) | 2.6 (0.40)
Statistical Analysis 1: Comparison: Asenapine vs Olanzapine; The null hypothesis was that there was no difference in change from baseline in body weight between asenapine and olanzapine at Day 182; Test type: Superiority or Other; p < 0.0001, Mixed Model for Repeated Measurements — [p-value comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded at each visit through end of treatment in this protocol (6 months). For subjects who did not continue in an extension protocol, serious adverse events (SAEs) were recorded via telephone 30 days after end of treatment.
Description: Information regarding AEs was obtained by questioning or examining the
  subject at each visit, and recording complaints and symptoms.
  Reports are for all SAEs and treatment-emergent nonserious AEs.
Arm/Group | Asenapine | Olanzapine
Serious Adverse Events (participants affected / at risk) | 30/244 | 18/224
Other Adverse Events (participants affected / at risk) | 145/244 | 140/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine (N=244) | Olanzapine (N=224)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Endocrine disorders) | 0 (0) | 1 (1)
VENTRICULAR EXTRASYSTOLES (General disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 1 (1)
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
PORCELAIN GALLBLADDER (Hepatobiliary disorders) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 1 (1)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
GRAND MAL CONVULSION (Nervous system disorders) | 1 (1) | 1 (1)
HEMORRHAGIC STROKE (Nervous system disorders) | 1 (1) | 0 (0)
ALCOHOL ABUSE (Psychiatric disorders) | 1 (1) | 0 (0)
HOMICIDAL IDEATION (Psychiatric disorders) | 1 (1) | 1 (1)
PSYCHOTIC DISORDER (Psychiatric disorders) | 4 (4) | 1 (1)
SCHIZOPHRENIA (Psychiatric disorders) | 11 (11) | 10 (11)
SCHIZOPHRENIA, PARANOID TYPE (Psychiatric disorders) | 8 (8) | 6 (6)
SCHIZOPHRENIA, UNDIFFERENTIATED TYPE (Psychiatric disorders) | 1 (1) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 4 (4) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine (N=244) | Olanzapine (N=224)
DRY MOUTH (Gastrointestinal disorders) | 9 (9) | 18 (20)
NAUSEA (Gastrointestinal disorders) | 20 (23) | 11 (12)
WEIGHT INCREASED (Investigations) | 23 (23) | 48 (51)
INCREASED APPETITE (Metabolism and nutrition disorders) | 8 (8) | 12 (16)
AKATHISIA (Nervous system disorders) | 22 (29) | 13 (16)
DIZZINESS (Nervous system disorders) | 18 (19) | 21 (26)
HEADACHE (Nervous system disorders) | 33 (40) | 23 (26)
SEDATION (Nervous system disorders) | 16 (17) | 17 (19)
SOMNOLENCE (Nervous system disorders) | 36 (38) | 43 (62)
ANXIETY (Psychiatric disorders) | 26 (37) | 16 (20)
INSOMNIA (Psychiatric disorders) | 43 (55) | 26 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Except for compelling legal reasons, neither the sponsor nor the investigator will communicate to third parties any result of the clinical trial before the clinical trial report has been released by the sponsor.